CLINICAL TRIAL: NCT00944450
Title: An Open-Label, Randomized, 2-Period, Single-Dose, Balanced, Crossover Study in Healthy Subjects to Establish the Bioequivalence of Tablet Formulations Containing the Anhydrous and Monohydrate (FMI) Forms of MK0431
Brief Title: Study of the Bioequivalence of Two Tablet Forms of MK0431 (0431-027)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0431-027; MK0431-027; 2009_614
Record Dates: First submitted 2009-07-21; First posted 2009-07-23 (Estimated); Results first posted 2010-04-27 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

ARMS (2):
- 1 (Active Comparator): Sitagliptin anhydrous formulation
  Interventions: Drug: Sitagliptin phosphate anhydrous formulation
- 2 (Active Comparator): Sitagliptin monohydrate FMI formulation
  Interventions: Drug: Comparator: sitagliptin phosphate monohydrate form

INTERVENTIONS:
Drug: Sitagliptin phosphate anhydrous formulation — Single dose sitagliptin 100 mg tablets (anhydrous form) in one of two treatment periods.
  Arms: 1
Drug: Comparator: sitagliptin phosphate monohydrate form — Single dose sitagliptin 100 mg tablets [monohydrate Final Market Image (FMI) form] in one of two treatment periods.
  Arms: 2

SUMMARY:
This study will establish that the MK0431 100 mg anhydrous formulation tablets are bioequivalent to the MK0431 100 mg monohydrate final market image (FMI) tablets.

ELIGIBILITY:
Inclusion Criteria:

* Subject is in good health
* Female subjects must have a negative pregnancy test
* Subject is within 30% of ideal body weight
* Subject does not smoke
* Subject agrees to follow the study guidelines

Exclusion Criteria:

* Subject has a history of any illness that might confound the results of the study or make participation unsafe for the subject
* Subject has a history of hypoglycemia
* Subject has a history of any hepatic disease
* Subject is taking any oral, parenteral, topical or implantable contraceptives

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2004-08; Primary Completion 2004-09 (Actual); Study Completion 2004-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Groups:
- 100 mg MK0431 Anhydrous Then 100 mg MK0431 Monohydrate: Single dose sitagliptin 100 mg tablets [monohydrate Final Market Image (FMI) form] in one of two treatment periods.
- 100 mg MK0431 Monohydrate Then 100 mg MK0431 Anhydrous: 100 mg MK0431 monohydrate (Phase III/FMI formulation) then 100 mg MK0431 anhydrous (Phase IIB formulation)
Period: Period 1
Arm/Group | 100 mg MK0431 Anhydrous Then 100 mg MK0431 Monohydrate | 100 mg MK0431 Monohydrate Then 100 mg MK0431 Anhydrous
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0
Period: Period 2
Arm/Group | 100 mg MK0431 Anhydrous Then 100 mg MK0431 Monohydrate | 100 mg MK0431 Monohydrate Then 100 mg MK0431 Anhydrous
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 12
Age, Continuous [Mean (Full Range); unit: years] | 45.3 [41 to 54]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 6
Height [Mean (Full Range); unit: Centimeters] | 170.5 [156.5 to 179.0]
Weight [Mean (Full Range); unit: Kilograms] | 75.3 [56.6 to 88.3]

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (AUC(0 to Infinity)) Following Single Dose Administration of the Anhydrous and Monohydrate Forms of MK0431 (Sitagliptin)
Description: Area Under the Plasma Concentration-Time Curve and peak concentration of the Anhydrous and Monohydrate Forms of MK0431 (Sitagliptin)
Time Frame: Through 72 Hours Following the Administration of the Medication
Population: Healthy Male and Female Subjects
Measure: Geometric Mean (Standard Deviation); unit: μmol*hr/L
Groups:
- 100 mg MK0431 Anhydrous: 100 mg MK0431 anhydrous (Phase IIB) formulation administered as a single dose.
- 100 mg MK0431 Monohydrate: 100 mg MK0431 monohydrate (Phase III/FMI) formulation administered as a single dose.
Arm/Group | 100 mg MK0431 Anhydrous | 100 mg MK0431 Monohydrate
Number analyzed (Participants) | 12 | 12
μmol*hr/L | 8.38 (0.77) | 8.78 (0.86)
Statistical Analysis 1: Comparison: 100 mg MK0431 Anhydrous vs 100 mg MK0431 Monohydrate; 100 mg MK0431 monohydrate (Phase III/FMI formulation) (B) vs. 100 mg MK0431 anhydrous (Phase IIB formulation) (A); Test type: Non-Inferiority or Equivalence — Pre-specified equivalence bounds = (0.80, 1.25) for AUC geometric mean ratio (B/A); Geometric Mean Ratio = 1.05, 90% CI [1.02 to 1.07]

2. Primary Outcome: Peak Plasma Concentration (Cmax) Following Single Dose Administration of the Anhydrous and Monohydrate Forms of MK0431 (Sitagliptin)
Description: Peak Plasma concentration (Cmax) for the Anhydrous and Monohydrate Forms of MK0431 (Sitagliptin)
Time Frame: Through 72 Hours Following the Administration of the Medication
Population: Healthy Male and Female Subjects
Measure: Geometric Mean (Standard Deviation); unit: μmol/L
Arm/Group | 100 mg MK0431 Anhydrous | 100 mg MK0431 Monohydrate
Number analyzed (Participants) | 12 | 12
μmol/L | 799 (164) | 856 (180)
Statistical Analysis 1: Comparison: 100 mg MK0431 Anhydrous vs 100 mg MK0431 Monohydrate; 100 mg MK0431 monohydrate (Phase III/FMI formulation) (B) vs. 100 mg MK0431 anhydrous (Phase IIB formulation) (A); Test type: Non-Inferiority or Equivalence — Pre-specified equivalence bounds = (0.80, 1.25) for Cmax geometric mean ratio (B/A); Geometric Mean Ratio = 1.07, 90% CI [0.94 to 1.22]

ADVERSE EVENTS:
Arm/Group | 100 mg MK0431 Anhydrous Then 100 mg MK0431 Monohydrate | 100 mg MK0431 Monohydrate Then 100 mg MK0431 Anhydrous
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 3/12 | 5/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 100 mg MK0431 Anhydrous Then 100 mg MK0431 Monohydrate (N=12) | 100 mg MK0431 Monohydrate Then 100 mg MK0431 Anhydrous (N=12)
Nausea (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1
Thermal Burn (Injury, poisoning and procedural complications) | 0 | 1
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.